CLINICAL TRIAL: NCT05763537
Title: Understanding the Role of Doulas in Supporting People With PMADs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 162-22
Record Dates: First submitted 2023-02-01; First posted 2023-03-10 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-06

CONDITIONS: Maternal Health; Pregnancy; Delivery, Obstetric; Self Efficacy; Social Support; Mental Health; Substance-Related Disorders; Postpartum Depression; Depression; Mental Health Services
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders; Depression, Postpartum; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Doula Care Plus the PMAD Intervention (Experimental): Participants in this arm will receive standard perinatal doula care provided by doulas trained in the DONA International doula training in addition to PMAD-specific care from their doulas.
  Interventions: Behavioral: Standard Doula Care Plus PMAD Intervention
- Standard Doula Care (Active Comparator): Participants in this arm will receive standard perinatal doula care provided by doulas trained in the DONA International doula training.
  Interventions: Behavioral: Standard Doula Care
- Standard Maternal Care (No Intervention): In this arm participants will receive standard perinatal medical care and will not receive care from a doula.

INTERVENTIONS:
Behavioral: Standard Doula Care Plus PMAD Intervention — Doulas trained in the DONA training, and the PMAD-focused training will provide care to perinatal people.
  Arms: Standard Doula Care Plus the PMAD Intervention
Behavioral: Standard Doula Care — Doulas trained in the DONA training will provide care to perinatal people.
  Arms: Standard Doula Care

SUMMARY:
Detailed Description The doula-led intervention developed during the first phase of this project will be pilot tested for feasibility. Following the recruitment procedures described in the recruitment and retention plan, approximately 75 participants will be enrolled into the study. Twenty-five of the participants will receive regular doula care and 25 of the participants will receive care from a doula trained in the PMAD doula training throughout their pregnancy, childbirth, and postpartum time period, following the intervention procedures developed in Aim 2 of this study. Twenty-five women will not receive care from a doula and will receive perinatal care as usual. Women in all groups will take surveys via REDCap during their enrollment in the intervention, at 1 month postpartum, 3 months, and 6 months postpartum (at the conclusion of the intervention). All participants who receive the PMAD doula intervention will complete checklists after each session with their doula, to assess fidelity to the intervention. Participant communication with their doula via patient notebook will also be assessed for fidelity to the intervention.

DETAILED DESCRIPTION:
Detailed Description The doula-led intervention developed during the first phase of this project will be pilot tested for feasibility. Following the recruitment procedures described in the recruitment and retention plan, approximately 75 participants will be enrolled into the study. Twenty-five of the participants will receive regular doula care and 25 of the participants will receive care from a doula trained in the PMAD doula training throughout their pregnancy, childbirth, and postpartum time period, following the intervention procedures developed in Aim 2 of this study. Twenty-five women will not receive care from a doula and will receive perinatal care as usual. Women in all groups will take surveys via REDCap during their enrollment in the intervention, at 1 month postpartum, 3 months, and 6 months postpartum (at the conclusion of the intervention). All participants who receive the PMAD doula intervention will complete checklists after each session with their doula, to assess fidelity to the intervention. Participant communication with their doula via patient notebook will also be assessed for fidelity to the intervention. A subsection of 20 participants who receive care from doulas in the PMAD training will also be eligible to participate in a qualitative interview at 6 months postpartum. The interview guide will be developed based on prior research with doulas, the PI's current research exploring doula-care in Montana, and feedback from the CAB. Example questions are expected to include: "What were your experiences working with a doula?" "What would have made your experience better?" and "What worked and what didn't work?"

Interviewers will all be graduate students who have completed research methods courses and will be trained by the PI, who has extensive experience in conducting qualitative research and in conducting qualitative interviews.

The following procedures will be followed:

1. Once participants have indicated that they are interested in participating in the study, the PI will contact them to set up a time to discuss the study with them, and if they are interested and meet eligibility criteria, enroll them in the study. Participants will be randomly assigned to either receive standard care from a doula, the doula PMAD intervention, or perinatal care as usual.
2. Before enrollment in the study, participants will be provided with a copy of the consent form, and the information on the consent form will be read to the participants.
3. Once the participants have provided informed consent, they will be given the pre-test survey via REDCap and will take the survey again at 1 month postpartum and 3 months postpartum.
4. All participants will be connected to a doula and receive either care as usual from a doula or a doula trained in the intervention by the PI and will engage in care with them throughout their pregnancy, during childbirth, and for 3 months postpartum. The exact components of the doula care provided will be developed in aim 2 based on the findings of study 1.
5. Participants will be provided compensation (in the form of a gift card) after the completion of each survey (pre-test, 1 month postpartum, 3 and 6 months postpartum).
6. At the completion of the study, participants will be thanked for their time and participation. For those who agreed to do member checks, participants will be re-contacted after analysis for member checks.

Participants who are randomized into the intervention arm of the study will also be randomly selected to participate in cross-sectional, semi-structured interviews.

Participant recruitment is described in the recruitment and retention plan. Participants will be interviewed about experience in the intervention.

The following steps will be followed:

1. Once participants have indicated that they are interested in participating in the interview portion of the study, the PI will contact them to set up a time for an interview and about their preferred interview site. They will have the option to do a phone interview if they are not available for an in-person interview or if they are not comfortable with an in-person interview for privacy reasons. The first interview will take place before they begin care with their doula.
2. Interview sessions will be scheduled at a pre-determined time at locations desired by the participants. If the interview takes place in person, Covid-19 protocols will be followed and include the completion of a Covid-19 symptom questionnaire by both the participant and the interviewer, the wearing of face masks during the interview, and social distancing.
3. Before beginning the interview, participants will be provided with a copy of the consent form, and the information on the consent form will be read to the participants. This process is further described in the Protection of Human Subjects document.
4. Once the participants have provided informed consent and provided consent to having the interview audio-recorded, the interviewer will begin recording the interview. A semi-structured interview guide will be used to guide the interview.
5. Audio-recorded interviews will follow semi-structured interview guides and last 60-90 minutes.
6. Following the interview, participants will be asked whether they are willing to be contacted to do a follow-up interview at 3 months postpartum.
7. Participants will be provided their compensation.
8. Participants will be thanked for their time and participation.
9. For those who agreed to do a second and third interviews at 3 and 6 months postpartum, the same process will be followed to conduct their second interview.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over the age of 18
* Currently pregnant and between 13 and 26 gestational weeks at the time of enrollment
* Live in a HRSA-designated rural area of Montana

Exclusion Criteria:

* They are under the age of 18
* Not currently pregnant
* Not between 13-26 gestational weeks at the time of enrollment
* If they do not live in a HRSA-designated rural are of Montana.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The Childbirth Self-Efficacy Inventory (CBSEI) | At study enrollment
  The Childbirth Self-Efficacy Inventory (CBSEI) is a 60-item self-report instrument that measures self-efficacy expectancies for coping with childbirth. In describing the development of the CBSEI, Lowe (1993) reports that the CBSEI scales have excellent internal consistency reliability (0.86 to 0.96) and factor analysis suggested that each CBSEl scale is unidimensional. Validity of the CBSEI was supported by significant positive correlations with the criterion variables of generalized self-efficacy, self-esteem, and internal health locus of control; and significant negative correlations with external health locus of control and learned helplessness. Validity was also supported by significantly higher self-efficacy scores for multiparous as compared to nulliparous pregnant women.
Change in the Childbirth Self-Efficacy Inventory (CBSEI) at 1 month postpartum | 1-month postpartum
  The Childbirth Self-Efficacy Inventory (CBSEI) is a 60-item self-report instrument that measures self-efficacy expectancies for coping with childbirth. In describing the development of the CBSEI, Lowe (1993) reports that the CBSEI scales have excellent internal consistency reliability (0.86 to 0.96) and factor analysis suggested that each CBSEl scale is unidimensional. Validity of the CBSEI was supported by significant positive correlations with the criterion variables of generalized self-efficacy, self-esteem, and internal health locus of control; and significant negative correlations with external health locus of control and learned helplessness. Validity was also supported by significantly higher self-efficacy scores for multiparous as compared to nulliparous pregnant women.
Change in the Childbirth Self-Efficacy Inventory (CBSEI) at 3 months postpartum | At 3-months
  The Childbirth Self-Efficacy Inventory (CBSEI) is a 60-item self-report instrument that measures self-efficacy expectancies for coping with childbirth. In describing the development of the CBSEI, Lowe (1993) reports that the CBSEI scales have excellent internal consistency reliability (0.86 to 0.96) and factor analysis suggested that each CBSEl scale is unidimensional. Validity of the CBSEI was supported by significant positive correlations with the criterion variables of generalized self-efficacy, self-esteem, and internal health locus of control; and significant negative correlations with external health locus of control and learned helplessness. Validity was also supported by significantly higher self-efficacy scores for multiparous as compared to nulliparous pregnant women.
Change in the Childbirth Self-Efficacy Inventory (CBSEI) at 6 months postpartum | At 6-months postpartum.
  The Childbirth Self-Efficacy Inventory (CBSEI) is a 60-item self-report instrument that measures self-efficacy expectancies for coping with childbirth. In describing the development of the CBSEI, Lowe (1993) reports that the CBSEI scales have excellent internal consistency reliability (0.86 to 0.96) and factor analysis suggested that each CBSEl scale is unidimensional. Validity of the CBSEI was supported by significant positive correlations with the criterion variables of generalized self-efficacy, self-esteem, and internal health locus of control; and significant negative correlations with external health locus of control and learned helplessness. Validity was also supported by significantly higher self-efficacy scores for multiparous as compared to nulliparous pregnant women.
The General Self-Efficacy Scale (SGSE) | At study enrollment
  The General Self-Efficacy Scale (SGSE) is a 17-item self-report instrument that measures perceived self-efficacy. Internal consistency reliability for the SGSE scale in organizational research has been moderate to high (alpha = .76 to .89) (e.g., Cable & Judge, 1994; Earley & Lituchy, 1991; Gardner & Pierce, 1998; Riggs & Knight, 1994; Schaubroeck & Merritt, 1997; Smith & Foti, 1998).
Change in the General Self-Efficacy Scale (SGSE) at 1-month postpartum | 1-month postpartum
  The General Self-Efficacy Scale (SGSE) is a 17-item self-report instrument that measures perceived self-efficacy. Internal consistency reliability for the SGSE scale in organizational research has been moderate to high (alpha = .76 to .89) (e.g., Cable & Judge, 1994; Earley & Lituchy, 1991; Gardner & Pierce, 1998; Riggs & Knight, 1994; Schaubroeck & Merritt, 1997; Smith & Foti, 1998).
Change in the General Self-Efficacy Scale (SGSE) at 3-months postpartum | At 3-months postpartum
  The General Self-Efficacy Scale (SGSE) is a 17-item self-report instrument that measures perceived self-efficacy. Internal consistency reliability for the SGSE scale in organizational research has been moderate to high (alpha = .76 to .89) (e.g., Cable & Judge, 1994; Earley & Lituchy, 1991; Gardner & Pierce, 1998; Riggs & Knight, 1994; Schaubroeck & Merritt, 1997; Smith & Foti, 1998).
Change in the General Self-Efficacy Scale (SGSE) at 6-months postpartum | At 6-months postpartum.
  The General Self-Efficacy Scale (SGSE) is a 17-item self-report instrument that measures perceived self-efficacy. Internal consistency reliability for the SGSE scale in organizational research has been moderate to high (alpha = .76 to .89) (e.g., Cable & Judge, 1994; Earley & Lituchy, 1991; Gardner & Pierce, 1998; Riggs & Knight, 1994; Schaubroeck & Merritt, 1997; Smith & Foti, 1998).
Edinburgh Depression Scale | At study enrollment
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report instrument that measures postnatal depression. A review of validation studies of the Edinburgh Depression Scale suggest the EPDS has high sensitivity and specificity (Eberhard-Gran et al., 2001). Other research supports its concurrent and predictive validity and Cronbach's alpha of between .82-.84 (Bergink et al., 2011).
Change in the Edinburgh Depression Scale at 1-month postpartum | At 1-month postpartum
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report instrument that measures postnatal depression. A review of validation studies of the Edinburgh Depression Scale suggest the EPDS has high sensitivity and specificity (Eberhard-Gran et al., 2001). Other research supports its concurrent and predictive validity and Cronbach's alpha of between .82-.84 (Bergink et al., 2011).
Change in the Edinburgh Depression Scale at 3-months postpartum | At 3-months postpartum.
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report instrument that measures postnatal depression. A review of validation studies of the Edinburgh Depression Scale suggest the EPDS has high sensitivity and specificity (Eberhard-Gran et al., 2001). Other research supports its concurrent and predictive validity and Cronbach's alpha of between .82-.84 (Bergink et al., 2011).
Change in Edinburgh Depression Scale at 6-months postpartum | At 6-months postpartum.
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report instrument that measures postnatal depression. A review of validation studies of the Edinburgh Depression Scale suggest the EPDS has high sensitivity and specificity (Eberhard-Gran et al., 2001). Other research supports its concurrent and predictive validity and Cronbach's alpha of between .82-.84 (Bergink et al., 2011).
Patient Health Questionnaire (PHQ)-9 | At study enrollment
  The Patient Health Questionnaire (PHQ)-9 is a 9-item self-report instrument that measures depression. The PHQ-9 has high criterion validity (.88 sensitivity, .88 specificity) and reliability of .86-.89 (Kroenke et al., 2021).
Change in Patient Health Questionnaire at 1-month postpartum (PHQ)-9 | At 1-month postpartum
  The Patient Health Questionnaire (PHQ)-9 is a 9-item self-report instrument that measures depression. The PHQ-9 has high criterion validity (.88 sensitivity, .88 specificity) and reliability of .86-.89 (Kroenke et al., 2021).
Change in Patient Health Questionnaire at 3-months postpartum (PHQ)-9 | At 3-months postpartum.
  The Patient Health Questionnaire (PHQ)-9 is a 9-item self-report instrument that measures depression. The PHQ-9 has high criterion validity (.88 sensitivity, .88 specificity) and reliability of .86-.89 (Kroenke et al., 2021).
Change in Patient Health Questionnaire at 6-months postpartum (PHQ)-9 | At 6-months postpartum.
  The Patient Health Questionnaire (PHQ)-9 is a 9-item self-report instrument that measures depression. The PHQ-9 has high criterion validity (.88 sensitivity, .88 specificity) and reliability of .86-.89 (Kroenke et al., 2021).
Generalized Anxiety Disorder (GAD)-7 | At study enrollment
  The GAD-7 screens for and is a symptom severity measure for four of the most common anxiety disorders. Spitzer et al.,(2006) describe strong support of the GAD-7: "Studies with the GAD indicate that the internal consistency of the GAD-7 is excellent (Cronbach α = .92). Test-retest reliability is also good (intraclass correlation = 0.83). Comparison of scores derived from the self-report scales with those derived from the MHP-administered versions of the same scales yielded similar results (intraclass correlation = 0.83), indicating good procedural validity. As the cut point increases, sensitivity decreases and specificity increases in a continuous fashion. At a cut point of 10 or greater, sensitivity and specificity exceed 0.80, and sensitivity is nearly maximized. The GAD-7 also has strong construct validity. There is a strong association between increasing GAD-7 severity scores and worsening function on all 6 SF-20 scales."
Change in Generalized Anxiety Disorder (GAD)-7 at 1-month postpartum | At 1-month postpartum
  The GAD-7 screens for and is a symptom severity measure for four of the most common anxiety disorders. Spitzer et al.,(2006) describe strong support of the GAD-7: "Studies with the GAD indicate that the internal consistency of the GAD-7 is excellent (Cronbach α = .92). Test-retest reliability is also good (intraclass correlation = 0.83). Comparison of scores derived from the self-report scales with those derived from the MHP-administered versions of the same scales yielded similar results (intraclass correlation = 0.83), indicating good procedural validity. As the cut point increases, sensitivity decreases and specificity increases in a continuous fashion. At a cut point of 10 or greater, sensitivity and specificity exceed 0.80, and sensitivity is nearly maximized. The GAD-7 also has strong construct validity. There is a strong association between increasing GAD-7 severity scores and worsening function on all 6 SF-20 scales."
Change in Generalized Anxiety Disorder (GAD)-7 at 3-months postpartum | At 3-months postpartum.
  The GAD-7 screens for and is a symptom severity measure for four of the most common anxiety disorders. Spitzer et al.,(2006) describe strong support of the GAD-7: "Studies with the GAD indicate that the internal consistency of the GAD-7 is excellent (Cronbach α = .92). Test-retest reliability is also good (intraclass correlation = 0.83). Comparison of scores derived from the self-report scales with those derived from the MHP-administered versions of the same scales yielded similar results (intraclass correlation = 0.83), indicating good procedural validity. As the cut point increases, sensitivity decreases and specificity increases in a continuous fashion. At a cut point of 10 or greater, sensitivity and specificity exceed 0.80, and sensitivity is nearly maximized. The GAD-7 also has strong construct validity. There is a strong association between increasing GAD-7 severity scores and worsening function on all 6 SF-20 scales."
Change in Generalized Anxiety Disorder (GAD)-7 at 6 months postpartum | At 6-months postpartum.
  The GAD-7 screens for and is a symptom severity measure for four of the most common anxiety disorders. Spitzer et al.,(2006) describe strong support of the GAD-7: "Studies with the GAD indicate that the internal consistency of the GAD-7 is excellent (Cronbach α = .92). Test-retest reliability is also good (intraclass correlation = 0.83). Comparison of scores derived from the self-report scales with those derived from the MHP-administered versions of the same scales yielded similar results (intraclass correlation = 0.83), indicating good procedural validity. As the cut point increases, sensitivity decreases and specificity increases in a continuous fashion. At a cut point of 10 or greater, sensitivity and specificity exceed 0.80, and sensitivity is nearly maximized. The GAD-7 also has strong construct validity. There is a strong association between increasing GAD-7 severity scores and worsening function on all 6 SF-20 scales."
Multi-Dimensional Scale of Perceived Social Support (MSPSS) | At study enrollment
  The MSPSS is a 12-item measure of perceived social support from three sources. Internal reliability of the MSPSS is strong using Cronbach's coefficient alphas (.91) (Dahlem et al., 1991).
Change in Multi-Dimensional Scale of Perceived Social Support (MSPSS) at 1-month postpartum | At 1-month postpartum
  The MSPSS is a 12-item measure of perceived social support from three sources. Internal reliability of the MSPSS is strong using Cronbach's coefficient alphas (.91) (Dahlem et al., 1991).
Change in Multi-Dimensional Scale of Perceived Social Support (MSPSS) at 3-months postpartum | At 3-months postpartum.
  The MSPSS is a 12-item measure of perceived social support from three sources. Internal reliability of the MSPSS is strong using Cronbach's coefficient alphas (.91) (Dahlem et al., 1991).
Change in Multi-Dimensional Scale of Perceived Social Support (MSPSS) at 6-months postpartum | At 6-months postpartum.
  The MSPSS is a 12-item measure of perceived social support from three sources. Internal reliability of the MSPSS is strong using Cronbach's coefficient alphas (.91) (Dahlem et al., 1991).
Social Support Questionnaire (SSQ)- Short Form | At study enrollment
  The SSQ-Short Form is a 6-item measure of social support that measures the number of people available to provide support in 6 different areas. The internal reliability of the short-version is high (.97-.98) (Sarason et al.,1987).
Change in Social Support Questionnaire (SSQ)- Short Form at 1-month postpartum | At 1-month postpartum
  The SSQ-Short Form is a 6-item measure of social support that measures the number of people available to provide support in 6 different areas. The internal reliability of the short-version is high (.97-.98) (Sarason et al.,1987).
Change in Social Support Questionnaire (SSQ)- Short Form at 3-months postpartum | At 3-months postpartum.
  The SSQ-Short Form is a 6-item measure of social support that measures the number of people available to provide support in 6 different areas. The internal reliability of the short-version is high (.97-.98) (Sarason et al.,1987).
Change in Social Support Questionnaire (SSQ)- Short Form at 6-months postpartum | At 6-months postpartum.
  The SSQ-Short Form is a 6-item measure of social support that measures the number of people available to provide support in 6 different areas. The internal reliability of the short-version is high (.97-.98) (Sarason et al.,1987).
Birth Companion Support Questionnaire | 1-month postpartum
  The BCSQ is comprised of 17-items to measure participants perception of lay birth companion support during labor. Research by Dunne et al., (2014) notes internal consistency (Cronbach's alpha is between .66-.76) and content and construct validity of the questionnaire (Dunne et al., 2014).
Change in Birth Companion Support Questionnaire at 3-months postpartum | At 3-months
  The BCSQ is comprised of 17-items to measure participants perception of lay birth companion support during labor. Research by Dunne et al., (2014) notes internal consistency (Cronbach's alpha is between .66-.76) and content and construct validity of the questionnaire (Dunne et al., 2014).
Change in Birth Companion Support Questionnaire at 6-months postpartum | At 6-months postpartum
  The BCSQ is comprised of 17-items to measure participants perception of lay birth companion support during labor. Research by Dunne et al., (2014) notes internal consistency (Cronbach's alpha is between .66-.76) and content and construct validity of the questionnaire (Dunne et al., 2014).
The Perceived Wellness Scale | At study enrollment
  The perceived wellness scale is a 36-item measure designed to assess an individual's own perception of their wellness through physical, spiritual,intellectual, psychological, social and emotional dimensions. Research by Adams (1995) indicates the scale has high factorial, discriminant, convergent and face validity. It also had high consistency (a = .91), and test-retest reliability (r = .73 to .81) (Adams, 1995).
Change in the Perceived Wellness Scale at 1-month postpartum | 1-month postpartum
  The perceived wellness scale is a 36-item measure designed to assess an individual's own perception of their wellness through physical, spiritual,intellectual, psychological, social and emotional dimensions. Research by Adams (1995) indicates the scale has high factorial, discriminant, convergent and face validity. It also had high consistency (a = .91), and test-retest reliability (r = .73 to .81) (Adams, 1995).
Change in the Perceived Wellness Scale at 3-months postpartum | 3-months postpartum
  The perceived wellness scale is a 36-item measure designed to assess an individual's own perception of their wellness through physical, spiritual,intellectual, psychological, social and emotional dimensions. Research by Adams (1995) indicates the scale has high factorial, discriminant, convergent and face validity. It also had high consistency (a = .91), and test-retest reliability (r = .73 to .81) (Adams, 1995).
Change in the Perceived Wellness Scale at 6-months postpartum | At 6-months postpartum.
  The perceived wellness scale is a 36-item measure designed to assess an individual's own perception of their wellness through physical, spiritual,intellectual, psychological, social and emotional dimensions. Research by Adams (1995) indicates the scale has high factorial, discriminant, convergent and face validity. It also had high consistency (a = .91), and test-retest reliability (r = .73 to .81) (Adams, 1995).
City Birth Trauma Scale City Birth Trauma Scale | At 1-month postpartum
  The City Birth Trauma Scale is a 29-item questionnaire developed to measure birth-related PTSD according to DSM-5 criteria of: stressor criteria (A), symptoms of re-experiencing (B), avoidance (C), negative cognitions and mood (D), and hyperarousal (E), as well as duration of symptoms (F), significant distress or impairment (E), and exclusion criteria or other causes (H). It has a high alpha of .92 (Ayers et al., 2018).
Change in the City Birth Trauma Scale at 3-months postpartum City Birth Trauma Scale | At 3-months postpartum
  The City Birth Trauma Scale is a 29-item questionnaire developed to measure birth-related PTSD according to DSM-5 criteria of: stressor criteria (A), symptoms of re-experiencing (B), avoidance (C), negative cognitions and mood (D), and hyperarousal (E), as well as duration of symptoms (F), significant distress or impairment (E), and exclusion criteria or other causes (H). It has a high alpha of .92 (Ayers et al., 2018).
Change in the City Birth Trauma Scale at 6-months postpartum City Birth Trauma Scale | At 6-months postpartum
  The City Birth Trauma Scale is a 29-item questionnaire developed to measure birth-related PTSD according to DSM-5 criteria of: stressor criteria (A), symptoms of re-experiencing (B), avoidance (C), negative cognitions and mood (D), and hyperarousal (E), as well as duration of symptoms (F), significant distress or impairment (E), and exclusion criteria or other causes (H). It has a high alpha of .92 (Ayers et al., 2018).

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) Alcohol Use Disorders Identification Test (AUDIT) | At study enrollment
  The Alcohol Use Disorders Identification Test(AUDIT) is a 10-item self-report measure that identifies alcohol consumption, drinking behaviors, and alcohol-related problems among adults. As described in a review by Reinert and Allen (2007): Over a broad range of diverse samples and settings the AUDIT has demonstrated a high degree of internal consistency. In a reliability generalization analysis of studies that appeared in 2000 or before, Shields and Caruso (2003) calculated a median reliability of 0.81, with a range of 0.59 to 0.91. Psychometric properties of the AUDIT, such as test-retest reliability and internal consistency, are high.
Change in the Alcohol Use Disorders Identification Test (AUDIT) at 1-month postpartum Alcohol Use Disorders Identification Test (AUDIT) | At 1-month postpartum
  The Alcohol Use Disorders Identification Test(AUDIT) is a 10-item self-report measure that identifies alcohol consumption, drinking behaviors, and alcohol-related problems among adults. As described in a review by Reinert and Allen (2007): Over a broad range of diverse samples and settings the AUDIT has demonstrated a high degree of internal consistency. In a reliability generalization analysis of studies that appeared in 2000 or before, Shields and Caruso (2003) calculated a median reliability of 0.81, with a range of 0.59 to 0.91. Psychometric properties of the AUDIT, such as test-retest reliability and internal consistency, are high.
Change in the Alcohol Use Disorders Identification Test (AUDIT) at 3-months postpartum Alcohol Use Disorders Identification Test (AUDIT) | 3-months postpartum
  The Alcohol Use Disorders Identification Test(AUDIT) is a 10-item self-report measure that identifies alcohol consumption, drinking behaviors, and alcohol-related problems among adults. As described in a review by Reinert and Allen (2007): Over a broad range of diverse samples and settings the AUDIT has demonstrated a high degree of internal consistency. In a reliability generalization analysis of studies that appeared in 2000 or before, Shields and Caruso (2003) calculated a median reliability of 0.81, with a range of 0.59 to 0.91. Psychometric properties of the AUDIT, such as test-retest reliability and internal consistency, are high.
Change in the Alcohol Use Disorders Identification Test (AUDIT) at 6-months postpartum Alcohol Use Disorders Identification Test (AUDIT) | At 6-months postpartum
  The Alcohol Use Disorders Identification Test(AUDIT) is a 10-item self-report measure that identifies alcohol consumption, drinking behaviors, and alcohol-related problems among adults. As described in a review by Reinert and Allen (2007): Over a broad range of diverse samples and settings the AUDIT has demonstrated a high degree of internal consistency. In a reliability generalization analysis of studies that appeared in 2000 or before, Shields and Caruso (2003) calculated a median reliability of 0.81, with a range of 0.59 to 0.91. Psychometric properties of the AUDIT, such as test-retest reliability and internal consistency, are high.
Drug Abuse Screening Test (DAST) | At study enrollment
  The Drug Abuse Screening Test (DAST) is a 10- item self-report form used to assess drug use with adults. The following evaluation of the scale is provided by Skinner (1982): The internal consistency reliability estimate was substantial at .92, and a factor analysis of item intercorrelations suggested an unidimensional scale. With respect to response style biases, the DAST was only moderately correlated with social desirability and denial. Concurrent validity was examined by correlating the DAST with background variables, frequency of drug use during the past 12 months, and indices of psychopathology.
Change in the Drug Abuse Screening Test (DAST) at 1-month postpartum | At 1-month postpartum
  The Drug Abuse Screening Test (DAST) is a 10- item self-report form used to assess drug use with adults. The following evaluation of the scale is provided by Skinner (1982): The internal consistency reliability estimate was substantial at .92, and a factor analysis of item intercorrelations suggested an unidimensional scale. With respect to response style biases, the DAST was only moderately correlated with social desirability and denial. Concurrent validity was examined by correlating the DAST with background variables, frequency of drug use during the past 12 months, and indices of psychopathology.
Change in the Drug Abuse Screening Test (DAST) at 3-months postpartum | At 3-months postpartum
  The Drug Abuse Screening Test (DAST) is a 10- item self-report form used to assess drug use with adults. The following evaluation of the scale is provided by Skinner (1982): The internal consistency reliability estimate was substantial at .92, and a factor analysis of item intercorrelations suggested an unidimensional scale. With respect to response style biases, the DAST was only moderately correlated with social desirability and denial. Concurrent validity was examined by correlating the DAST with background variables, frequency of drug use during the past 12 months, and indices of psychopathology.
Change in the Drug Abuse Screening Test (DAST) at 6-months postpartum | At 6-months postpartum.
  The Drug Abuse Screening Test (DAST) is a 10- item self-report form used to assess drug use with adults. The following evaluation of the scale is provided by Skinner (1982): The internal consistency reliability estimate was substantial at .92, and a factor analysis of item intercorrelations suggested an unidimensional scale. With respect to response style biases, the DAST was only moderately correlated with social desirability and denial. Concurrent validity was examined by correlating the DAST with background variables, frequency of drug use during the past 12 months, and indices of psychopathology.
CDC Health-Related Quality of Life (HRQOL)- 4 scale | At study enrollment
  The CDC Health-Related Quality of Life (HRQOL)-4 is a 4-item self-report measure of personal health and wellbeing. A large body of research indicates the HRQOL's construct and criterion validity (CDC, 2000) and high retest reliability (.75 or higher) (Andresen et al., 2003).
Change in the CDC Health-Related Quality of Life (HRQOL)- 4 scale at 1-month postpartum | At 1-month postpartum
  The CDC Health-Related Quality of Life (HRQOL)-4 is a 4-item self-report measure of personal health and wellbeing. A large body of research indicates the HRQOL's construct and criterion validity (CDC, 2000) and high retest reliability (.75 or higher) (Andresen et al., 2003).
Change in the CDC Health-Related Quality of Life (HRQOL)- 4 scale at 3-months postpartum | At 3-months postpartum.
  The CDC Health-Related Quality of Life (HRQOL)-4 is a 4-item self-report measure of personal health and wellbeing. A large body of research indicates the HRQOL's construct and criterion validity (CDC, 2000) and high retest reliability (.75 or higher) (Andresen et al., 2003).
Change in the CDC Health-Related Quality of Life (HRQOL)- 4 scale at 6-months postpartum | At 6-months postpartum
  The CDC Health-Related Quality of Life (HRQOL)-4 is a 4-item self-report measure of personal health and wellbeing. A large body of research indicates the HRQOL's construct and criterion validity (CDC, 2000) and high retest reliability (.75 or higher) (Andresen et al., 2003).
Pregnancy Risk Assessment Monitoring (PRAMS) | 1 time during the study period, at 1-month postpartum.
  The core PRAMS questionnaire is a 52-item survey asking questions about behaviors and experiences during pregnancy, labor and the postpartum time period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Montana, Missoula, Montana, United States